CLINICAL TRIAL: NCT02166541
Title: Evaluation of "Intensive Neurophysiological Rehabilitation System" (INRS) With "Biomechanical Correction of the Spine According to Kozyavkin" (BCSK) in Children With Spastic Bilateral Cerebral Palsy: a Randomized Controlled Trial.
Brief Title: Evaluation of INRS With BCSK in Children With Spastic Bilateral Cerebral Palsy: a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: International Clinic of Rehabilitation, Ukraine (Other)
Responsible Party: Principal Investigator, Hans Forssberg, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Forssberg_KI_1
Record Dates: First submitted 2014-06-09; First posted 2014-06-18 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Spastic Diplegia Cerebral Palsy
Keywords: cerebral palsy, spastic, diplegic,; children,; intervention study,; manipulation, spinal; randomized controlled trial
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- INRS with BCSK (Experimental): "Intensive Neurophysiological Rehabilitation System (INRS)" including the "Biomechanical correction of the spine according to Kozyavkin (BCSK)".
  The daily treatment for about 2 hours are in general equal for all children except for the type of spinal manipulation. Duration of all treatment will be noted in a Treatment Diary.
  Interventions: Procedure: BCSK; Procedure: INRS
- INRS with traditional spinal manipulation (Sham Comparator): "Intensive Neurophysiological Rehabilitation System (INRS)" including spinal manipulation by the traditional technique.
  The daily treatment for about 2 hours are in general equal for all children except for the type of spinal manipulation. Duration of all treatment will be noted in a Treatment Diary.
  Interventions: Procedure: Traditional spinal manipulation; Procedure: INRS
- Total population (Experimental): All participants (i.e., both arms described above INRS with BCSK or traditional spinal manipulation)
  Interventions: Procedure: BCSK; Procedure: Traditional spinal manipulation; Procedure: INRS

INTERVENTIONS:
Procedure: BCSK — The "BCSK" is a specific technique of polysegmental spinal manipulation developed by Professor Kozyavkin based on applying quick short impulse aimed on moving intervertebral joints outside restrictive barrier.
  Arms: INRS with BCSK; Total population
Procedure: Traditional spinal manipulation — Spinal manipulation by traditional technique is a mild mobilization without impulse, based on applying gentle repetitive force without crossing restrictive barrier.
  Arms: INRS with traditional spinal manipulation; Total population
Procedure: INRS — The "INRS" is a treatment program developed at the International Clinic of Rehabilitation where the spinal manipulation is one of several components. There may be some variation in treatment depending on the clinical situation. All children receive the main treatment components which are massage, physical therapy, warm wax and paraffin applications and low electro stimulation with a special portable device as a part of treatment called "Reflexotherapy".

SUMMARY:
A randomized control trial investigating "Biomechanical Correction of the Spine according to Kozyavkin" (BCSK) which is a part of the treatment concept "Intensive Neurophysiological Rehabilitation System" (INRS). BCSK is used with the aims to reduce muscle tone and improve gross and fine motor function in children with Spastic Bilateral Cerebral Palsy.

DETAILED DESCRIPTION:
The study is a collaboration between the International Clinic of Rehabilitation (ICR) in Ukraine and the Karolinska Institute (KI) in Sweden. The intervention and the assessments are performed at ICR. The primary outcome measure, evaluation of gross motor function with the test GMFM 66 is filmed and the recordings are transferred to KI together with all assessment data. KI are responsible for study research design and collects, analyzes and processes all data. It is a double blinded study. Only two persons will know to which group the subject belongs, the person performing the randomization process in Sweden and the doctor performing the spinal corrections.

There are two aims of the study;

1. To evaluate the effect of "Biomechanical Correction of the Spine" (BCSK) in children with Spastic Bilateral Cerebral Palsy.
2. To evaluate the effect of "Intensive Neurophysiological Rehabilitation System" (INRS) in children with Spastic Bilateral Cerebral Palsy.

ELIGIBILITY:
Inclusion criteria:

* Children with Spastic Bilateral form of Cerebral Palsy according Surveillance of Cerebral Palsy in Europe (SCPE) criteria
* GMFCS levels II-IV
* The children should not have received previous INRS treatment

Exclusion Criteria:

* Other forms of Cerebral Palsy
* Severe epileptic syndrome
* Severe mental retardation
* Orthopedic surgery within the last year

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure 66 (GMFM 66) is used to measure change over time | Baseline, 2 weeks, 6 months
  The Gross Motor Function Measure (GMFM) evaluates gross motor function in children with cerebral palsy. This version, GMFM 66, contains 66 items that span the spectrum from activities in lying and rolling up to walking, running and jumping skills.

SECONDARY OUTCOMES:
Muscle tone testing using Modified Ashworth Scale is used to measure change over time | Baseline, 2 weeks, 6 months
  Estimation of muscle tone during rapid passive extension of the tested muscle-groups according to an ordinal scale.

OTHER OUTCOMES:
Box and Blocks test is used to measure change over time | Baseline, 2 weeks, 6 months
  Evaluation of fine motor skills using Box and Blocks test. The score is the number of blocks carried from one compartment to the other in one minute. Each hand is scored separately.
Range of motion is used to measure change over time | Baseline, 2 weeks, 6 months
  Range of motion measurement with goniometer in wrist, elbow, hip, knee and ankle joints.
Boyd and Graham´s Selective Motor Control Scale is used to measure change over time | Baseline, 2 weeks, 6 months
  Performance of voluntary active ankle dorsiflexion according the ordinal scale, Boyd and Graham´s Selective Motor Control Scale.
NeuroFlexor is used to measure change over time | Baseline, 2 weeks, 6 months
  Testing of muscle tone using the NeuroFlexor when applicable. The NeuroFlexor (Aggero MedTech AB, Solna, Sweden) is an instrument for objectively quantifying passive movement in wrist and finger flexor muscles.
Questionnaire is used to measure change over time | 2 weeks, 6 months
  Questionnaire of treatment efficiency, filled in by parents.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Forssberg, Professor, Principal Investigator — Department of Women´s and Children´s Health, Karolinska University
Locations (1):
- International Clinic of Rehabilitation, Truskavets, Lviv Oblast, Ukraine